CLINICAL TRIAL: NCT06681259
Title: Clinical Specialty Queue For Gestational Trophoblastic Neoplasia
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weiguo Lv, Doctor, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: IRB-20240344-R
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gestational Trophoblastic Neoplasia
MeSH Terms: conditions — Gestational Trophoblastic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to establish a bidirectional cohort study of GTN specific diseases, including 1020 retrospective cases Queue and 1000 prospective cohorts. Based on the clinical collaboration system for gynecological tumors in multiple tertiary hospitals across the country, establish unified criteria for case inclusion and exclusion, and establish a multi center clinical queue for GTN; Collect baseline information of GTN patients, such as age, reproductive history, environmental and social information, genetic related information, physical examination, physicochemical, imaging, and pathological information; Collect biological specimens such as blood/tissue from patients; Collect information related to the diagnosis, treatment plan, human chorionic gonadotropin (hCG) levels, and toxic side effects of patients during the diagnosis and treatment period; After the end of treatment, follow-up blood hCG levels, imaging, fertility status, as well as recurrence and metastasis status, are conducted to track prognosis, thus building a clinical diagnosis and treatment information database, forming a standardized follow-up system for GTN, identifying high-risk factors for GTN chemotherapy resistance, constructing a precise evaluation model for GTN resistance, and providing high-level evidence-based medicine for effectively improving the initial treatment efficacy of GTN.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥ 18 years old; ② Patients clinically diagnosed with GTN (including invasive cases) Molar pregnancy, choriocarcinoma, PSTT, ETT); ③ Complete informed consent for enrollment.

Exclusion Criteria:

* ① Having mental illness or cognitive impairment, unable to cooperate in completing the investigation with Patients with concurrent malignant tumors; ③ Participants with severe missing follow-up data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collaborate with multiple tertiary hospitals nationwide to collect ethical approvals for gynecological oncology clinical trials and include them in the group Information on GTN patients who received treatment at participating units within the next 5 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2029-11-04 (Estimated); Study Completion 2029-11-04 (Estimated)

PRIMARY OUTCOMES:
Collect disease-related clinical and pathological features of the included subjects | GTN should be closely followed up after treatment, with monthly follow-up once in the first year and 2-3 days Follow up once every 3 months annually for a total of 5 years.
  Collect baseline information of GTN patients, such as age, reproductive history,environmental and social information, genetic related information, physical examination, physicochemical, imaging, and pathological information; Collect biological specimens such as blood/tissue from patients; Collect information on the diagnosis, treatment plan, levels of human chorionic gonadotropin, and toxic side effects of patients during the diagnosis and treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Weiguo Lv, Zhengjiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No